CLINICAL TRIAL: NCT07165613
Title: Do Different Taping Methods Enhance Performance in Adolescent Volleyball Players With Patient-Reported Ankle Instability?
Brief Title: Effects of Taping on Performance in Adolescent Volleyball Players With Patient-Reported Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Feyza Sule BADILLI HANTAL, Asst.Prof, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: taping
Record Dates: First submitted 2025-08-30; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Functional Ankle Instability
Keywords: Ankle; ankle injuries; physical functional performance; athletic tape
MeSH Terms: conditions — Ankle Injuries | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiotaping (Experimental): Kinesiotape is applied
  Interventions: Other: Kinesiotape
- Dynamic tape (Experimental): dynamic tape applied
  Interventions: Other: Dynamic tape
- control (No Intervention): no intervention

INTERVENTIONS:
Other: Kinesiotape — Kinesiotape is applied
  Arms: Kinesiotaping
Other: Dynamic tape — dynamic tape applied
  Arms: Dynamic tape

SUMMARY:
The purpose of this study is to investigate the effects of different types of taping application to functional performancein adolescent volleyball players with functional ankle instability. The Cumberland Ankle Instability Tool was used to select participants, 27 and less than 27 scores were included. Twenty-nine players mean age is 13,49±2,1 were included. Functional performance tests (Single Leg Hop Test, Triple Hop Test, Crossover Hop Test, 6 m. Hop Time Test) were applied to all players according to results control group and taping groups ( kinesiology tape group, dynamic tape group ) were created. Immediately, functional performance test were repeated after kinesiology taping and dynamic taping applied. Statistically no significant difference was found between control groups and both taping groups (p>0,05). When the results of taping and non-taping compared, significant difference was not found (p>0,05). As a result, we may say that taping has no effect to functional performance on players with functional ankle instability. More study is needed about effects of taping to functional performance on athletes with sports injuries.

ELIGIBILITY:
inclusion criteria: Athletes scoring 27 or below active volleyball players without recent severe lower extremity injuries exclusion criteria: having surgery within six months, ankle injuries in the preceding month. Those scoring above 27, having recent injuries, surgery, or metabolic disorders

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Single Leg Hop Test | Baseline (Pre-taping): Immediately before taping Post-intervention (Post-taping): Immediately after taping
  Single Leg Hop Test
Triple hop test | Baseline (Pre-taping): Immediately before taping Post-intervention (Post-taping): Immediately after taping
  Triple hop test
crossover hop test | Baseline (Pre-taping): Immediately before taping Post-intervention (Post-taping): Immediately after taping
  crossover hop test
6m timed hop test | Baseline (Pre-taping): Immediately before taping Post-intervention (Post-taping): Immediately after taping
  6m timed hop test

SECONDARY OUTCOMES:
t scores | Baseline (Pre-taping): Immediately before taping Post-intervention (Post-taping): Immediately after taping
  t scores

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Sule Badilli Hantal, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: thesis — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- Available data/document: thesis — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp